CLINICAL TRIAL: NCT03342352
Title: A Randomized, Global, Phase 3 Trial of Nivolumab Plus Epacadostat in Combination With Chemotherapy (Platinum + 5-fluorouracil) Versus the EXTREME Regimen (Cetuximab + Platinum + 5-fluorouracil) in First-line Treatment of Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN) / CheckMate 9NA /ECHO-310
Brief Title: Nivolumab Plus Epacadostat in Combination With Chemotherapy Versus the EXTREME Regimen in Squamous Cell Carcinoma of the Head and Neck (CheckMate 9NA/ECHO-310)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was cancelled prior to enrolling any patients.
Sponsor: Incyte Corporation (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA2099NA/ECHO-310
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Head and Neck Cancer
Keywords: Squamous cell carcinoma of the head and neck; programmed cell death protein 1 (PD-1) antibody; indoleamine 2,3-dioxygenase (IDO) inhibitor
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Nivolumab; epacadostat; Carboplatin; Cisplatin; Cetuximab; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Nivolumab plus epacadostat in combination with platinum (carboplatin/cisplatin) plus 5-fluorouracil.
  Interventions: Drug: Nivolumab; Drug: Epacadostat; Drug: Carboplatin; Drug: Cisplatin; Drug: 5-Fluorouracil
- Arm B (Active Comparator): EXTREME regimen.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Cetuximab; Drug: 5-Fluorouracil
- Arm C (Experimental): Nivolumab plus placebo for epacadostat in combination with platinum (carboplatin/cisplatin) plus 5-fluorouracil.
  Interventions: Drug: Nivolumab; Drug: Placebo; Drug: Carboplatin; Drug: Cisplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Nivolumab — Nivolumab administered intravenously at the protocol-defined dose every 3 weeks.
  Arms: Arm A; Arm C
Drug: Epacadostat — Epacadostat administered orally at the protocol-defined dose twice daily.
  Other Names: INCB024360
  Arms: Arm A
Drug: Placebo — Matching placebo for epacadostat administered orally twice daily.
  Arms: Arm C
Drug: Carboplatin — Carboplatin administered intravenously at the protocol-defined dose every 3 weeks for 6 cycles.
Drug: Cisplatin — Cisplatin administered intravenously at the protocol-defined dose every 3 weeks for 6 cycles.
Drug: Cetuximab — Cetuximab administered intravenously at the protocol-defined dose weekly.
  Arms: Arm B
Drug: 5-Fluorouracil — 5-Fluorouracil administered intravenously at the protocol-defined dose on Days 1-4 for 6 cycles.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the combination of nivolumab plus epacadostat in combination with chemotherapy in first-line recurrent or metastatic patients with squamous cell carcinoma of the head and neck (SCCHN) when compared to the standard of care (EXTREME regimen).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed SCCHN from any of the following primary sites: oral cavity, oropharynx, hypopharynx, and larynx.
* Must have recurrent or metastatic disease that is not amenable to therapy with curative intent (surgery and/or radiation therapy with or without chemotherapy).
* No prior treatment with systemic anti-cancer therapy for SCCHN unless protocol-defined conditions are met.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to1.
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST v1.1.
* Documentation of program death ligand-1 (PD-L1) status prior to randomization.

Exclusion Criteria:

* Recurrent or metastatic carcinoma of the nasopharynx and paranasal sinuses, squamous cell carcinoma that originated from the skin and salivary gland or non-squamous histologies (e.g., mucosal melanoma) and SCCHN of unknown primary origin.
* Untreated central nervous system (CNS) metastases.
* Carcinomatous meningitis.
* Active, known or suspected autoimmune disease.
* Physical and laboratory test findings outside the protocol-defined range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) with nivolumab plus epacadostat in combination with chemotherapy (Arm A) compared to the EXTREME regimen (Arm B) | Up to approximately 35 months
  Defined as the time between the date of randomization and the date of first documented disease progression (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1]) or death due to any cause, whichever occurs first.
Overall survival (OS) with nivolumab plus epacadostat in combination with chemotherapy (Arm A) compared to the EXTREME regimen (Arm B) | Up to approximately 48 months
  Defined as the time between the date of randomization and the date of death.

SECONDARY OUTCOMES:
Objective response rate (ORR) with nivolumab plus epacadostat in combination with chemotherapy (Arm A) and the EXTREME regimen (Arm B) | Up to approximately 35 months
  Defined as the number of participants with a best overall response of complete response (CR) or partial response (PR) divided by the number of randomized participants for each treatment group.
Duration of response (DOR) with nivolumab plus epacadostat in combination with chemotherapy (Arm A) and the EXTREME regimen (Arm B) | Up to approximately 35 months
  Defined as the time between the date of first documented response (CR or PR per RECIST v1.1) to the date of the first disease progression (per RECIST v1.1) or death due to any cause, whichever occurs first.
ORR with nivolumab plus placebo in combination with chemotherapy (Arm C) | Up to approximately 35 months
  Defined as the number of participants with a best overall response of complete response (CR) or partial response (PR) divided by the number of randomized participants for each treatment group.
PFS with nivolumab plus placebo in combination with chemotherapy (Arm C) | Up to approximately 35 months
  Defined as the time between the date of randomization and the date of first documented disease progression (per RECIST v1.1) or death due to any cause, whichever occurs first.
DOR with nivolumab plus placebo in combination with chemotherapy (Arm C) | Up to approximately 35 months
  Defined as the time between the date of first documented response (CR or PR per RECIST v1.1) to the date of the first disease progression (per RECIST v1.1) or death due to any cause, whichever occurs first.
Time to meaningful symptomatic deterioration (TTSD) with nivolumab plus epacadostat in combination with chemotherapy (Arm A) compared to the EXTREME regimen (Arm B) | Up to approximately 60 months
  TTSD assessed by the 10-item Functional Assessment of Cancer Therapy-Head & Neck (FACT-HN) Symptom Index (FHNSI-10).

CONTACTS AND LOCATIONS:
Overall Officials: Vinny Hayreh, MD, Study Director — Bristol-Myers Squibb Research and Development

IPD SHARING:
Plan to Share IPD: No